

## STATISTICAL ANALYSIS PLAN FOR PART 1 USING PROTOCOL AMTX100-AD-01

**Sponsor:** 

amytrx

Amytrx Therapeutics, Inc.

**Protocol Number:** AMTX100-AD-01 (NCT04313400)

**Protocol Title:** A Two part, Phase I/II, Multi-center, Double-Blind,

Randomized, Vehicle-controlled Study of the Safety and Efficacy of topically applied AMTX-100 CF in adult patients

with Mild to Moderate Atopic Dermatitis

**Protocol Version / Date:** Final Version 2.0/20 Jan 2020

**SAP Author:** Amarex Clinical Research,

LLC

20201 Century Boulevard

Germantown, MD 20874

USA

1-

Telephone:

1-866-AMAREX-1 1-301-528-7000

Facsimile: 1-301-528-2300

**Plan Version:** Part 1 Version 1.0

Plan Date: 16Sep2021

| Protocol Number: | AMTX100-AD-01 |
|---|---|
| <b>Protocol Version / Date:</b> | Final Version 2.0/ 20 Jan 2020 |
| Protocol Name: | A Two part, Phase I/II, Multi-center, Double-Blind, Randomized, Vehicle-controlled Study of the Safety and Efficacy of topically applied AMTX-100 CF in adult patients with Mild to Moderate Atopic |
| Sponsor: | Amytrx Therapeutics, Inc. |
| Prepared by: | Amarex Clinical Research<br>20201 Century Boulevard<br>Germantown, Maryland 20874 |
| SAP Version: | Part 1 Version 1.0 |
| SAP Date: | 16Sep2021 |
| I have read and approve the Statistics Statistician, Amarex Clinical Res | ical Analysis Plan specified above and agree on its content: search Date |
| SPONSOR Representative | Date |

## TABLE OF CONTENTS

| Section | on | | Page |
|---|---|---|---|
| ABB | REVIAT | IONS, ACRONYMS, AND DEFINITIONS | 5 |
| 1. | INTE | CODUCTION | 7 |
| 2. | PRO | PROTOCOL DESIGN | |
| | 2.1 | Design Overview | |
| | 2.2 | Cohorts | |
| | 2.3 | Randomization and Stratification | |
| | 2.4 | Blinding | |
| | 2.5 | Protocol Objective(s) | 12 |
| | 2.6 | Secondary Objective | |
| | 2.6 | Efficacy Assessments/ Outcome Measures | |
| 3. | | PLE SIZE DETERMINATION, STATISTICAL POWER, AND SIGNIFIC | |
| 4. | | RIM ANALYSIS | |
| 5. | PRIN | ARY HYPOTHESIS TO BE TESTED | 13 |
| 6. | ANA | LYSIS POPULATIONS | 14 |
| | 6.1 | Safety Population | 14 |
| 7. | DAT | A CONVENTION AND RELATED DEFINITIONS | 14 |
| | 7.1 | Baseline Definition | 14 |
| | 7.2 | Duplicate Data | |
| | 7.3 | Outliers | |
| | 7.4 | Handling of Missing Data | |
| | 7.5 | Multicenter Clinical Trials | |
| | 7.6 | Multiple Comparisons and Multiplicity | |
| | 7.7 | Covariates and Prognostic Factors | |
| | 7.8 | Subgroups | |
| | 7.9 | Standard Calculations | 15 |
| | | 7.9.1 Age | |
| | | 7.9.2 Change from baseline | |
| | | 7.9.3 Percent Change from Baseline | |
| 8. | | TISTICAL METHODS | |
| | 8.1 | Summarizing Disposition and Baseline Data | |
| | | 8.1.1 Subject Disposition and Withdrawals | |
| | | 8.1.3 Demographics and Baseline Characteristics | |
| | | 8.1.4 Prior and Concomitant Medications | |
| | | 8.1.5 Extent of Exposure | |
| | | 8.1.6 Study Treatment Compliance | |
| | 8.2 | Analysis of Safety Data | |
| | | 8.2.1 Adverse Events | |
| | | 8.2.3 Clinical Laboratory Evaluations | |
| | | 8.2.4 Vital Signs | |
| | | 8.2.5 Physical Examination | |

| | | 8.2.6 | Urine Pregnancy Test | 20 |
|-----|------|---------|-----------------------|----|
| 9. | APPE | NDIX 1. | | 21 |
| 10. | APPE | NDIX 2 | | 23 |
| | 10.1 | Planne | d by-subject listings | 23 |
| | 10.2 | Planne | d Summary Tables | 24 |
| 11. | REFE | RENCES | 5 | 25 |
| 12. | VERS | ION HIS | TORY | 26 |

## ABBREVIATIONS, ACRONYMS, AND DEFINITIONS

Abbreviation/Acronym Definition

AD Atopic Dermatitis

AE Adverse Event

ANCOVA Analysis of Covariance

ASA American Statistical Association

BMI Body Mass Index

BP Blood Pressure

BSA Body Surface Area

CI Confidence Interval

CM Concomitant Medications

CRF Case Report Form

CRO Contract Research Organization

CTCAE Common Terminology Criteria for Adverse Events

DLQI Dermatology Life Quality Index

DLT Dose-Limiting Toxicity

DSMC Data Safety Monitoring Committee

EASI Eczema Area and Severity Index

eCRF Electronic Case Report Form

FDA U.S. Food and Drug Administration

IA Interim Analysis

ICF Informed Consent Form

ICH International Council on Harmonization

IDMC Independent Data Monitoring Committee

ITT Intent-to-Treat

IWRS Interactive Web Randomization System

MedDRA Medical Dictionary for Regulatory Activities

MTD Maximum Tolerable Dose

NRS Pruritus Numerical Rating Scale

PI Principal Investigator

PT Preferred Term level of MedDRA

QOL On Quality of Life

Protocol: AMTX100-AD-01 Amytrx Therapeutics, Inc.

| Abbreviation/Acronym | <b>Definition</b> |
|---|---|
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| $SAS^{	ext{	ext{$\mathbb{R}$}}}$ | Statistical Analysis System |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| TCS | Topical corticosterioids |
| TEAE | Treatment-emergent Adverse Event |
| USA | United States of America |
| vIGA-AD | Validated Investigator Global Assessment for Atopic Dermatitis |
| WHO | World Health Organization |

#### 1. INTRODUCTION

This Statistical Analysis Plan describes the planned analyses and reporting for the Phase I (Part 1) clinical trial protocol AMTX100-AD-01, conducted by Amytrx Therapeutics, Inc. The reader of this Statistical Analysis Plan (SAP) is encouraged to review the complete protocol and amendments as this plan contains only a limited overview of protocol information. The main objectives of this plan are to provide details pertaining to statistical methodology, data conventions, and processes used for the analysis of data from this trial.

The format and content of this SAP are structured to provide sufficient detail to meet the requirements specified by the International Council on Harmonization (ICH) E9: Guidance on Statistical Principles in Clinical Trials. All work planned and presented in this Statistical Analysis Plan will follow the ethical guidelines published by the American Statistical Association (ASA).

The following documents were reviewed in preparation of this Statistical Analysis Plan:

- Final protocol 2.0/ 20 Jan 2020
- ASA Ethical Guidelines for Statistical Practice (2016)
- The Royal Statistical Society: Code of Conduct (2014)
- ICH Guidance on the Structure and Content of Clinical Study Reports (ICH E3, 1996)
- ICH Guidance on the Structure and Content of Clinical Study Reports (ICH E3(R1), 2013)
- ICH Guidance on the Statistical Principles for Clinical Trials (ICH E9, 1998)
- ICH Guidance on the Statistical Principles for Clinical Trials (ICH E9(R1), 2017)

#### 2. PROTOCOL DESIGN

#### 2.1 Design Overview

This is an adaptive, Phase I study: Part 1 (Maximum Tolerable Dose (MTD) Finding by maximum percentage of BSA treated).

Part 1 of this study is an open-label, dose escalation study of the safety and tolerability of topically applied AMTX-100 CF in adult patients with mild to moderate AD. Part I of this study is designed to determine the MTD of AMTX-100 CF (1.1% w/w concentration) for the highest treated percentage of the BSA affected with AD. The MTD is defined as 1 cohort dose level below the dose, in which dose limiting toxicities (DLTs) as defined below were observed. In total, five (5) cohort dose levels will be tested sequentially by escalating applications of AMTX-100 CF 1.1% to higher percentages of BSA affected with AD at each cohort. Each enrolled subject will receive the assigned dose of Open-label AMTX-100 CF 1.1% w/w to be applied twice daily to all treatable lesions of AD

Protocol: AMTX100-AD-01 Amytrx Therapeutics, Inc.

(excluding the scalp, face, eyes, eyelids, neck, hands, palms, feet, groin, genitals or in the axillae) for 7 consecutive days (14 applications in total), regardless of whether the lesions become clinically clear during the 7 day treatment period.



Assuming no DLTs occur at any cohorts, in Part 2 (Phase II) of the study, three dose concentrations (low doset-treatment safety. concentration (0.11% w/w), medium dose concentration (0.33% w/w) and high dose concentration (1.1% w/w)) of AMTX-100 CF will be further evaluated for safety and efficacy, compared to placebo (vehicle), in adult patients with mild to moderate AD, with up to 70% treatable BSA involvement.



#### 2.2 Cohorts

The cohorts to be evaluated in this study described as Table 2-1.



#### 2.3 Randomization and Stratification

There is no randomization for the Phase I (Part 1) of the study.

## 2.4 Blinding

There is no blinding for the Phase I (Part 1) of the study.

## 2.5 Protocol Objective(s)

## **Primary Objective**

 To determine the MTD of topically applied AMTX-100 CF (in 1.1% w/w concentration) in adult patients with mild to moderate Atopic Dermatitis (AD) while escalating the treatable BSA involved in sequential cohorts.

#### **Secondary Objective**

• To evaluate the safety, tolerability and efficacy of topically applied AMTX-100 CF (in 1.1%

w/w concentration) in improving symptoms associated with mild to moderate Atopic Dermatitis in adults.

## 2.6 Efficacy Assessments/ Outcome Measures

## 2.6.1.1 Primary Outcome Measure

 Maximum Tolerable Dose (MTD) by maximum percentage of BSA treated, by evaluation of dose-limiting toxicity (DLT) of AMTX-100 CF (1.1% w/w concentration) based on the safety profile

## 2.6.1.2 Safety Outcome Measures

- Incidence of Treatment-Emergent Adverse Events (TEAE)
- Incidence of withdrawals from the study due to TEAEs
- Changes in study treatment application site reaction assessment
- Changes and shifts in laboratory measurements over time
- Changes in vital signs over time

# 3. Sample Size Determination, Statistical Power, And Significance Level

The sample size of 25 subjects (5 subjects per cohort) for Phase I of this study is selected on the basis of clinical judgment and not based on statistical power calculation. The number of subjects is deemed adequate to provide clinically meaningful descriptive results consistent with study objectives.

| 4. | INTERIM ANALYSIS | C | , , |
|----|------------------|---|-----|

#### 5. PRIMARY HYPOTHESIS TO BE TESTED

There is no formal hypothesis testing for this study as the study is a Phase I evaluation and is not intended to be hypothesis generating. The study is not powered to reliably yield statistically significant conclusions.

| 6. | ANALYSIS POPULATIONS |
|---|---|
| 7. | DATA CONVENTION AND RELATED DEFINITIONS |
| 7.4 | Handling of Missing Data |
| All eff | forts will be made to avoid missing data; however there will be no imputation of missing data |
| for thi | s early phase study and all summaries will be based on observed data only |
| 7.5 | Multicenter Clinical Trials |
| This is | s a multi-center clinical trial. |

# 7.8 Subgroups

There is no prespecified subgroup analysis for this study. Subgroup analysis may be conducted as needed.





## 8. STATISTICAL METHODS

All statistical analyses will be performed using SAS® for Windows, version 9.4 or later. All data collected during this study will be presented in subject data listings.



# 8.1 Summarizing Disposition and Baseline Data

## 8.1.1 Subject Disposition and Withdrawals

There will be a detailed accounting of all subjects who sign an informed consent to participate in this trial. The following will be summarized by cohort:



#### **8.1.2** Protocol Deviations

Protocol deviations for all randomized subjects will be listed as by-subject listing and deviations will be summarized descriptively according to the following categories:



## 8.1.3 Demographics and Baseline Characteristics

Demographics and baseline characteristics (including age, race, gender, Ethnicity, Height, Weight, BMI and BSA etc.) will be presented as by-subject listing and summarized by cohort.

Atopic dermatitis history and medical history will be provided as by-subject listings.

#### **8.1.4** Prior and Concomitant Medications

Prior medication is defined as any medications with an end date prior to the first treatment date.

All prior and concomitant medications recorded in the case report form will be listed and coded to the drug substance level (i.e., generic term) using the most recent version of WHO Drug dictionary, and summarized by cohort and by the number and percentage of subjects taking each medication for the Safety population.

## 8.1.5 Extent of Exposure

All treatment administration data will be listed and summarized for the Safety population.

The extent of exposure will be summarized descriptively.

| 8.1.6 S | Study Treatment Compliance |
|---------|----------------------------|

# 8.2 Analysis of Safety Data

All safety analyses will be conducted using the Safety population. All data collected will be summarized according to the variable type. No inferential statistics are planned.

#### 8.2.1 Adverse Events

Adverse events will be classified by system organ class (SOC) and preferred term (PT) according to the most recent version of MedDRA dictionary.

TEAE are defined as adverse events with onset date on or after the first treatment. TEAEs will be summarized by cohort, System Organ Class, and preferred term. The following TEAE summaries will be provided:



All adverse events recorded in the eCRF will be presented as by-subject listings.

#### **8.2.2** Application Site Reaction

Local skin reactions will be assessed in all areas treated with study drug and graded by the investigator on a scale of 0 to 4 based on the area with the most severe skin reaction among all treated areas. A grade of 0 represents no reaction, and a grade of 4 indicates a marked and severe skin reaction that extended beyond the treated areas.

| I |
|---|

## 8.2.3 Clinical Laboratory Evaluations

All results of laboratory evaluations will be presented as by-subject listings. 8.2.4 Vital Signs Vital sign assessments are performed in order to characterize basic body function. The parameters collected in this study are: systolic BP (mmHg), diastolic BP (mmHg), temperature (<sup>0</sup>C), heart rate (bpm), respiratory rate (bpm).

| 8.2.5 Physical Examination |
|----------------------------|

| 8.2.6 Urine Pregnancy Test |
|---|
| All data from Urine Pregnancy test will be presented as a by-subject listing. |

## 9. APPENDIX 1

FIGURE 9-1: PHASE I (PART 1) - SCHEDULE OF ASSESSMENTS

| | | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 |
|---|---|---|---|---|---|---|
| Visit | | (Screening) | (Phone call) | (Baseline) | (End of | (Follow Up) |
| | | | | | Treatment) | |
| Days From Randomization | | Up to -21 days | Up to -7 days | Day 0 | Day +7 | Day +21 |
| Weeks From Randomization | | Week -3 | Week -1 | Week 0 | Week 1 | Week 3 |
| Window Period | | | ±2 days | | | ±2 days |
| | Protocol Section | | | | | |
| | | X | | | | |
| | | X | X | | | |
| | | X | | | | |
| | | X | | | | |
| | | X | | $X^{[1]}$ | | |
| | | X | | $X^{[1]}$ | X | X |
| | | X | | | | |
| | | X | | $X^{[1]}$ | X | X |
| | | X | | $X^{[1]}$ | X | X |
| | | X | | $X^{[1]}$ | X | X |
| | | X | | X <sup>[1]</sup> | X | X |
| | | X | | X <sup>[1]</sup> | X | |
| | | | | X <sup>[1]</sup> | X | X |

| X | | X <sup>[1]</sup> | X | X |
|---|---|------------------------------------------|---|---|
| | X | | | |
| | | X | | |
| | | X | | |
| | | 2 <sup>nd</sup> dose (PM) on Day 0, then | | |
| | | BID through Day 6 | | |
| | | $X^{[2]}$ | X | |
| | | | X | |
| | | X <sup>[1][2]</sup> | X | X |
| | | X <sup>[2]</sup> | X | X |

#### 10. APPENDIX 2



# **10.2 Planned Summary Tables**



#### 11. REFERENCES

- 1. ASA Ethical Guidelines for Statistical Practice (2016)
- 2. The Royal Statistical Society: Code of Conduct (2014)
- 3. ICH Guidance on the Structure and Content of Clinical Study Reports (ICH E3, 1996)
- 4. ICH Guidance on the Structure and Content of Clinical Study Reports (ICH E3(R1), 2013)
- 5. ICH Guidance on the Statistical Principles for Clinical Trials (ICH E9, 1998)
- 6. ICH Guidance on the Statistical Principles for Clinical Trials (ICH E9(R1), 2017)
- 7. Badia X, Mascaro JM, et al. Measuring health-related quality of life in patients with mild to moderate eczema and psoriasis: clinical validity, reliability and sensitivity to change of the DLQI. Br J Dermatol 1999; 141:698-702.
- 8. Basra MK, Salek MS, Camilleri L, Sturkey R, Finlay AY. Determining the Minimal Clinically Important Difference and Responsiveness of the Dermatology Life Quality Index (DLQI): Further Data. Dermatology. 2015;230(1):27-33.
- Eli Lilly and Company. Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD<sup>TM</sup>). International Eczema Council 2017; http://www.eczemacouncil.org/wp-content/uploads/2018/02/Validated-Investigator-Global-Assessment-Scale vIGA-AD 2017.pdf

# 12. VERSION HISTORY

# Version 1

This is the first version of this document.